CLINICAL TRIAL: NCT00619086
Title: Does a Single Dose of Steroid Before Thyroidectomy Improve Postoperative Nausea, Pain and Vocal Function?
Brief Title: Steroid Before Thyroidectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bern (Other)
Responsible Party: Candinas Daniel, MD, Department of Visceral- and Transplantation Surgery
Allocation: Randomized | Model: Parallel | Masking: Triple
Other Study IDs: KEK_49_05
Record Dates: First submitted 2008-02-07; First posted 2008-02-20 (Estimated); Last update posted 2008-06-09 (Estimated); Status verified 2008-06

CONDITIONS: Thyroid Surgery for Benign Disease
Keywords: thyroidectomy; dexamethasone; steroid; nausea
MeSH Terms: conditions — Nausea

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- A, 1 (Placebo Comparator): Placebo 45 minutes prior to surgery
  Interventions: Drug: Placebo
- A, 2 (Active Comparator): 8 mg Dexamethasone 45 minutes prior to surgery
  Interventions: Drug: Dexamethason Helvepharm ®

INTERVENTIONS:
Drug: Dexamethason Helvepharm ® — 8 mg Dexamethason i.v. 45 minutes prior to surgery
  Arms: A, 2
Drug: Placebo — 100 ml sodium chloride i.v. 45 minutes prior to surgery
  Arms: A, 1

SUMMARY:
We evaluated the effects of giving a single dose of steroid before thyroid surgery in a single institutional, double-blinded, randomized controlled trial. Postoperative nausea, pain, and vocal function were significantly improved after steroid administration compared to controls.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing thyroid surgery for benign disease

Exclusion Criteria:

* Depression
* Chronic pain disorder
* Insulin dependent diabetes mellitus
* History of PONV
* Pregnancy
* Age < 18 years
* Received antiemetic therapy within 48 hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2005-11; Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Nausea | 0-72 hours postoperative

SECONDARY OUTCOMES:
Pain, vocal function | 0-72 hours postoperative

CONTACTS AND LOCATIONS:
Overall Officials: Stephan A. Vorburger, MD, Principal Investigator — Dept of visceral- and transplant surgery, University Hospital Bern
Locations (1):
- Department of visceral- and transplant surgery, Bern, Switzerland

REFERENCES:
- [Derived] Worni M, Schudel HH, Seifert E, Inglin R, Hagemann M, Vorburger SA, Candinas D. Randomized controlled trial on single dose steroid before thyroidectomy for benign disease to improve postoperative nausea, pain, and vocal function. Ann Surg. 2008 Dec;248(6):1060-6. doi: 10.1097/SLA.0b013e31818c709a. PMID 19092351